CLINICAL TRIAL: NCT07210190
Title: A Prospective Clinical Study Evaluating the Effects of a Topical Multivitamin Serum, Containing PDRN on Facial Skin Hydration and Biophysical Parameters Following Microneedling
Brief Title: Microneedling for Skin Heath
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Erevna Innovations Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO-2025-VAMP-02
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Aesthetic
Keywords: Topical; Polydeoxyribonucleotide; Skin booster; Skin; Hydration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - biweekly treatment schedule (Active Comparator): Participants in this group will undergo an initial microneedeling session followed by a topical application of standardized, non-crosslinked hyaluronic acid. Following this initial treatment participants in Group A will receive three treatments of microneedeling immediately followed by topical application of VAMP™ Topical Multivitamin Serum every two (2) weeks
  Interventions: Device: Microneedeling with topical application of VAMP™ Topical Multivitamin Serum
- Group B - month treatment schedule (Active Comparator): Participants in this group will undergo an initial microneedeling session followed by a topical application of standardized, non-crosslinked hyaluronic acid. Following this initial treatment participants in Group B will receive three treatments of microneedeling immediately followed by topical application of VAMP™ Topical Multivitamin Serum every four (4) weeks
  Interventions: Device: Microneedeling with topical application of VAMP™ Topical Multivitamin Serum

INTERVENTIONS:
Device: Microneedeling with topical application of VAMP™ Topical Multivitamin Serum — VAMP™ Topical Multivitamin Serum is not indicated for use in pregnancy, lactation, or in individuals under the age of 22. Female participants of childbearing potential will be required to undergo urine pregnancy testing at baseline and prior to each treatment session. They will also be instructed to use an acceptable form of effective contraception for the duration of the study.

SUMMARY:
Skin boosters are treatments designed to improve skin quality and restore skin health. Some of these treatments are based on polynucleotides, which are small fragments of DNA. One such compound, called Polydeoxyribonucleotide (PDRN), is obtained from fish sources such as salmon or trout. PDRN has shown regenerative and anti-inflammatory properties, and in medical practice it has been used to support wound healing, scar improvement, and skin rejuvenation by helping with elasticity, texture, and fine lines.

VAMP™ Multivitamin Serum is a topical formulation that contains PDRN along with amino acids, vitamins, and peptides. It is designed to improve hydration, elasticity, and overall skin radiance. While early data suggest potential benefits, clinical research is still limited, and further study is needed.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to adequately understand the verbal explanations and the written participant information provided in local language and ability and willingness to give consent to participate in the study. Signed and dated informed consent to participate in the study.
2. Participant interested in improving skin quality.
3. Immune-competent adult 22 years of age and older.
4. Has intent to undergo treatment to improve appearance of the facial skin.
5. Willingness to comply with pre-visit instructions, including shaving of facial area (for male participants), to allow for consistent biometric and photographic evaluations.
6. If the participant is a female of childbearing potential, she agrees to use an acceptable form of effective birth control for the duration of the study and is willing to take a urine pregnancy test (UPT) at Baseline and prior to receiving any study treatment.

   Acceptable forms of effective birth control include:
   * Barrier methods of contraception: Condom or occlusive cap (diaphragm or cervical caps) with spermicidal foam/gel/film/ cream/suppository;
   * Bilateral tubal ligation;
   * Combined oral contraceptives (estrogens and progesterone), implanted or injectable contraceptives on a stable dose for at least 28 days prior to Day 1;
   * Hormonal or copper intra uterine device (IUD) inserted at least 28 days prior to Day 1;
   * Vasectomized partner (in monogamous relationship) for at least 3 months prior to screening;
   * Strict abstinence (at least one month prior to baseline and agrees to continue for the duration of the study or use acceptable form of birth control).
7. Negative UPT for women of childbearing potential at the Baseline visit.
8. Stable lifestyle and skincare regimen for at least 4 weeks

Exclusion Criteria:1. Known or suspected allergy or hypersensitivity to any components of VAMP™ ADVANCED Topical Multivitamin Serum, including sodium hyaluronate, peptides, polynucleotides (e.g., PDRN), or excipients.

2. Known allergy or intolerance to topical anesthetics or lidocaine. 3. History of hypersensitivity reactions such as anaphylaxis, angioedema, or other severe allergic responses.

4. History of hypertrophic scarring, keloid formation, or post-inflammatory hyperpigmentation following cosmetic treatments.

5. Tattoos, piercings, or skin bleaching agents in the treatment area that may interfere with assessments, as judged by the Investigator.

6. Participants with known pigmentary instability or history of adverse response to microneedling.

7. Previous cosmetic or dermatologic procedures in the treatment area within the following time frames: 8. Previous treatment with cross-linked hyaluronic acid dermal fillers in the treatment area within the last 12 months.

9. Energy-based devices (laser, IPL, RF, ultrasound) in the last 6 months. 10. Microneedling, dermabrasion, mesotherapy, or chemical peels in the last 6 months.

11. Use of topical corticosteroids, retinoids, or depigmenting agents in the treatment area within the past 4 weeks.

12. Current use of immunosuppressive therapy, systemic corticosteroids, or chemotherapy within the last 3 months.

13. History of systemic autoimmune, collagen vascular, or bleeding disorders (e.g., lupus, scleroderma, thrombocytopenia).

14. Current pregnancy, positive urine pregnancy test at screening, breastfeeding, or intent to become pregnant during the study.

15. Participation in another clinical study within the past 30 days or concurrent participation in another interventional trial.

16. Any condition, including psychological, cognitive, or behavioral concerns, that would interfere with the ability to give informed consent, follow the protocol, or comply with follow-up requirements.

17. Initiation of a weight loss program or GLP-1 agonist therapy within 30 days before baseline or planned during study period.

18. Active skin conditions exacerbated by microneedling or transepidermal delivery, including chronic dermatitis or impaired barrier function.

19. Current participation by study personnel, immediate family members, or employees of the Sponsor.

20. Known allergy to fish or seafood, including but not limited to salmon, due to the potential presence of PDRN derived from marine sources.

21. History of cancer or previous radiation near or on the area to be treated. 22. Heavy smokers, classified as smoking more than 12 cigarettes per day. 23. Presence of any disease or lesions near or on the area to be treated, e.g.

1. Inflammation, active or chronic infection in or near the treatment area
2. Psoriasis, eczema, herpes zoster and acanthosis
3. Cancer or precancerous condition (e.g. actinic keratosis)
4. Severe skin laxity, flaccidity, or sagging
5. Advanced photoaged/ photodamaged skin (e.g., advanced skin elastosis, multiple lentigo solaris lesions) or skin condition (e.g., very crinkled, very thin, fragile skin or severe skin atrophy) in the treatment area that in the Investigator's opinion could interfere with the safety or effectiveness of the study product or injection procedure.

   24. Skin coloring/bleaching/tattoo in the treatment area, which, in the Treating Investigator's opinion, would interfere with the study injections and/or study assessment.

   25. An underlying known disease, a surgical or medical condition that would expose the participant to undue risk, e.g. history of bleeding disorders, active hepatitis, active autoimmune disease such as connective tissue diseases, systemic lupus erythematosus, polymyositis, dermatomyositis, multiple sclerosis or scleroderma.

   26. Use of concomitant medication that have the potential to prolong bleeding times such as anticoagulants or inhibitors of platelet aggregation (e.g., warfarin, clopidogrel, aspirin, baby aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs), Omega 3 or Vitamin E), within 14 days prior to injection. Omega 3 and Vitamin E are acceptable only as part of a standard Topical Multivitamin formulation. Cyclooxygenase-2 (COX 2) inhibitors are allowed.

   27. Treatment with chemotherapy, immunosuppressive agents, systemic corticosteroids within 3 months before treatment (inhaled or ophthalmic corticosteroids are allowed).

   28. Use of hormonal therapy (ex. HRT or contraceptives) unless the participant has been on a stable dose for at least 3 months prior to screening and does not plan to make any changes to the HRT regimen during the study period.

   29. Use of topical corticosteroids, topical prescription retinoids in the treatment area within 1 month of the Baseline visit or systemic retinoid treatment within 6 months of the baseline visit, or plan to receive such treatment.

   30. Pregnancy (confirmed by positive urine pregnancy test (UPT)/ serum pregnancy test), breast feeding or intends to become pregnant over the duration of the study.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-17 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Skin Hydration From Baseline | Baseline to final follow-up (Week 10 for Group A; Week 16 for Group B)
  Percentage change in skin hydration from Baseline following microneedling with sequential applications of VAMP™ Topical Multivitamin Serum, measured using the Corneometer CM 825 (Courage+Khazaka electronic GmbH).

SECONDARY OUTCOMES:
Change in Transepidermal Water Loss (TEWL) From Baseline | Baseline to final follow-up (Week 10 for Group A; Week 16 for Group B)
  Percentage change in TEWL from Baseline, measured using the Tewameter TM 21
Change in Skin Surface Biophysical Parameters From Baseline | Baseline to final follow-up (Week 10 for Group A; Week 16 for Group B)
  Percentage change in surface evaluation of living skin cells (SELS: roughness, scaliness, smoothness, desquamation, and pore size), measured via the VisioScan VC 98.
Change in Skin Elasticity From Baseline | Baseline to final follow-up (Week 10 for Group A; Week 16 for Group B)
  Percentage change in skin elasticity from Baseline, measured using the Cutometer Dual MPA 580.
Participant Satisfaction With Treatment | Week 2 to Week 10 for Group A; Baseline to Week 16 for Group B
  Proportion of participants who report being at least "satisfied" (satisfied, very much satisfied, or extremely satisfied) on a seven-point participant satisfaction scale
Global Aesthetic Improvement Scale (GAIS) Score Assessed by Blinded Evaluator | Baseline to Week 10 for Group A; Baseline to Week 16 for Group B
  Proportion of participants rated as "improved" (improved, much improved, or very much improved) on the GAIS by a blinded evaluator at the end of the study
Safety and Tolerability of Treatment | Baseline to final follow-up (Week 10 for Group A; Week 16 for Group B)
  Incidence and frequency of adverse events
Change in VISIA® CR Facial Imaging Metrics | Baseline to final follow-up (Week 10 for Group A; Week 16 for Group B)
  Percentage change from Baseline in VISIA® CR-derived facial metrics as assessed by non invasive analysis of facial images

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Nikolis, MD, PhD, Principal Investigator — Erevna Innovations Inc.
Locations (1):
- Erevna Innovations Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No